CLINICAL TRIAL: NCT06383910
Title: The Effect Of Square Stepping Exercise Training On Cognitive Functions And Quality Of Life In Geriatric Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Yelda Soykurt, Physiotherapist, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10.185.1.58
Record Dates: First submitted 2024-02-15; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: geriatric; cognitive functions; square stepping exercise; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The group which doesn't get any intervention.
- Exercise Group (Active Comparator): The group received square stepping exercise training three times a week for six weeks.
  Interventions: Behavioral: Square Stepping Exercise

INTERVENTIONS:
Behavioral: Square Stepping Exercise — The exercise is performed on a thin exercise mat divided into 40 small squares. Participants are shown specific step patterns on this mat and are instructed to repeat the same step pattern until the end of the exercise mat. Once a pattern is completed on the exercise mat, its mirror-image pattern is also performed. The basic pattern is repeated 3-5 times, followed by the same number of repetitions for the mirror-image pattern. However, if participants struggle with the pattern, it is repeated until they learn it. Individuals execute the demonstrated pattern on the exercise mat and return to the beginning of the mat after completing it.
  Arms: Exercise Group

SUMMARY:
This study was designed to investigate the effects of Square-Stepping Exercise Training on cognitive functions and quality of life in geriatric individuals. The volunteer participants in the study were randomly divided into two groups: a square-stepping exercise group and a control group.

In the study, participants in the exercise training groups received square stepping exercises three days a week for six weeks, while those in the control group did not undergo any training. Both groups were assessed before and six weeks after the training period.

The investigators used several assessment tools including Hodkinson's Mental Test, Montreal Cognitive Assessment, Stroop Test, Trail Making Test, and the Turkish World Health Organization Quality-of-Life Scale.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 65-75 years old,
* Able to walk independently,
* Hodkinson Mental Test score ≥ 8,
* Without any neurological or lower extremity-affecting diseases,
* Healthy geriatric individuals who agreed to participate in the study were included.

Exclusion Criteria:

* Using 3 or more medications,
* Hodkinson Mental Test score <8,
* Currently participating in any exercise/rehabilitation program,
* Geriatric individuals with a history of lower extremity surgery

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Change on Cognitive Functions from Base on the Montreal Cognitive Assessment In 6 Weeks | Baseline and 6 weeks
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
Change on Cognitive Functions from Base on the Stroop Test In 6 Weeks | Baseline and 6 weeks
  The Stroop test measures the interference between reading and naming the ink color of words, highlighting the conflict between automatic and controlled cognitive processes.
Change on Cognitive Functions from Base on the Trail Making Test In 6 Weeks | Baseline and 6 weeks
  The Trail Making Test is a test that involves visual scanning and working memory. Test consists of two parts, A and B. In Part A (TMT-A), the participant must draw a line to connect consecutive numbers, from 1 to 25. In Part B (TMT-B), the participant connects numbers and letters in an alternating progressive sequence, 1 to A, A to 2, 2 to B, and so on
Change on Quality of Live from Base on the World Health Organization Quality-of-Life Scale Turkish version In 6 Weeks | Baseline and 6 weeks
  The WHOQOL-OLD is an instrument for the assessment of subjective quality of life in elderly people.

CONTACTS AND LOCATIONS:
Overall Officials: Yelda Soykurt, Principal Investigator — PhD student
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)